CLINICAL TRIAL: NCT02303821
Title: Phase 1b/2 Study of Carfilzomib in Combination With Induction Chemotherapy in Children With Relapsed or Refractory Acute Lymphoblastic Leukemia
Brief Title: Study of Carfilzomib in Combination With Induction Chemotherapy in Children With Relapsed or Refractory Acute Lymphoblastic Leukemia
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Amgen (Industry)
Collaborators: Therapeutic Advances in Childhood Leukemia & Lymphoma (TACL) - Study Design & Execution Collaborator (Unknown); Innovative Therapies For Children with Cancer Consortium (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CFZ008; 2014-001633-84 (EudraCT Number)
Record Dates: First submitted 2014-11-20; First posted 2014-12-01 (Estimated); Results first posted 2025-06-04 (Actual); Last update posted 2025-06-04 (Actual); Status verified 2025-05

CONDITIONS: Acute Lymphoblastic Leukemia (ALL)
MeSH Terms: conditions — Precursor Cell Lymphoblastic Leukemia-Lymphoma | interventions — carfilzomib; WW Domain-Containing Oxidoreductase; Dexamethasone; Mitoxantrone; pegaspargase; Vincristine; Methotrexate; Hydrocortisone; Mercaptopurine; Cyclophosphamide; Cytarabine; Daunorubicin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Phase 1b: Dose Escalation 1 (Experimental): Subjects will receive carfilzomib in combination with induction chemotherapy, comprising an R3 backbone of dexamethasone, mitoxantrone, PEG asparaginase, and vincristine.
  Subjects will have a 1 week carfilzomib single agent Lead in Window prior to the Induction Cycle.
  Subjects will receive a 4 week cycle of induction chemotherapy and have the option to receive a 4 week cycle of consolidation chemotherapy (Children's Oncology Group (COG) modified Berlin Frankfurt Münster (BFM) chemotherapy backbone (6 mercaptopurine, cyclophosphamide, cytarabine, PEG asparaginase, vincristine), if stable disease or better response is achieved at the end of the Induction Cycle.
  Interventions: Drug: Carfilzomib; Drug: Dexamethasone; Drug: Mitoxantrone; Drug: PEG-asparaginase; Drug: Vincristine; Drug: Intrathecal (IT) Methotrexate; Drug: Intrathecal Triple Therapy (Intrathecal Cytarabine, Hydrocortisone, and Methotrexate); Drug: 6-Mercaptopurine; Drug: Cyclophosphamide; Drug: Cytarabine
- Phase 1b: Dose Escalation 2 (Experimental): Subjects will receive carfilzomib in combination with induction chemotherapy, comprising a VXLD backbone of vincristine, dexamethasone, PEG asparaginase, and daunorubicin.
  Subjects will receive a 4 week cycle of carfilzomib and induction chemotherapy and then have the option to receive a 4 week cycle of consolidation chemotherapy (Children's Oncology Group (COG) modified Berlin Frankfurt Münster (BFM) chemotherapy backbone (6 mercaptopurine, cyclophosphamide, cytarabine, PEG asparaginase, vincristine), if stable disease or better response is achieved at the end of the Induction Cycle.
  Interventions: Drug: Carfilzomib; Drug: Dexamethasone; Drug: PEG-asparaginase; Drug: Vincristine; Drug: Intrathecal (IT) Methotrexate; Drug: Intrathecal Triple Therapy (Intrathecal Cytarabine, Hydrocortisone, and Methotrexate); Drug: 6-Mercaptopurine; Drug: Cyclophosphamide; Drug: Cytarabine; Drug: Daunorubicin
- Phase 2: Aged ≥ 12 months at screening (Experimental): All subjects aged ≥ 12 months at screening.
  Subjects will receive the recommended phase 2 dose (RP2D) of carfilzomib determined in Phase 1b.
  Subjects will receive a 4 week cycle of carfilzomib and induction chemotherapy comprising of a VXLD backbone of vincristine, dexamethasone, PEG asparaginase and daunorubicin. Subjects will then have the option to receive a 4 week cycle of carfilzomib in combination with consolidation chemotherapy Children's Oncology Group (COG) modified Berlin Frankfurt Münster (BFM) chemotherapy backbone (6 mercaptopurine, cyclophosphamide, cytarabine, PEG asparaginase, vincristine) if subjects showed no disease progression at the end of the Induction Cycle.
  Interventions: Drug: Carfilzomib; Drug: Dexamethasone; Drug: PEG-asparaginase; Drug: Vincristine; Drug: Intrathecal (IT) Methotrexate; Drug: Intrathecal Triple Therapy (Intrathecal Cytarabine, Hydrocortisone, and Methotrexate); Drug: 6-Mercaptopurine; Drug: Cyclophosphamide; Drug: Cytarabine; Drug: Daunorubicin
- Phase 2: Aged < 12 months at screening (Experimental): All subjects aged < 12 months at screening.
  Subjects will receive the recommended phase 2 dose (RP2D) of carfilzomib determined in Phase 1b.
  Subjects will receive a modified 5 week cycle (based on Interfant-06) of carfilzomib and induction chemotherapy comprising of a VXLD backbone of vincristine, dexamethasone, PEG asparaginase and daunorubicin. Subjects will then have the option to receive a 5 week cycle (modified based on Interfant-06) of carfilzomib in combination with consolidation chemotherapy Children's Oncology Group (COG) modified Berlin Frankfurt Münster (BFM) chemotherapy backbone (6 mercaptopurine, cyclophosphamide, cytarabine, PEG asparaginase, vincristine), if subjects showed no disease progression at the end of the Induction Cycle.
  Interventions: Drug: Carfilzomib; Drug: Dexamethasone; Drug: PEG-asparaginase; Drug: Vincristine; Drug: Intrathecal (IT) Methotrexate; Drug: Intrathecal Triple Therapy (Intrathecal Cytarabine, Hydrocortisone, and Methotrexate); Drug: 6-Mercaptopurine; Drug: Cyclophosphamide; Drug: Cytarabine; Drug: Daunorubicin

INTERVENTIONS:
Drug: Carfilzomib
  Other Names: PR-171; PR171; Kyprolis® (carfilzomib) for Injection
Drug: Dexamethasone
Drug: Mitoxantrone
  Arms: Phase 1b: Dose Escalation 1
Drug: PEG-asparaginase
Drug: Vincristine
Drug: Intrathecal (IT) Methotrexate
Drug: Intrathecal Triple Therapy (Intrathecal Cytarabine, Hydrocortisone, and Methotrexate)
Drug: 6-Mercaptopurine
Drug: Cyclophosphamide
Drug: Cytarabine
Drug: Daunorubicin
  Arms: Phase 1b: Dose Escalation 2; Phase 2: Aged < 12 months at screening; Phase 2: Aged ≥ 12 months at screening

SUMMARY:
The purpose of Phase 1b of this study is to:

* Asses the safety, tolerability and activity of carfilzomib, alone and in combination with induction chemotherapy, in children with relapsed or refractory acute lymphoblastic leukemia (ALL).
* Determine the maximum tolerated dose (MTD) and to recommend a phase 2 dose of carfilzomib in combination with induction chemotherapy.

The purpose of Phase 2 of this study is to compare the rate of complete remission (CR) of carfilzomib in combination with vincristine, dexamethasone, PEG asparaginase, daunorubicin (VXLD) at the end of induction therapy to an appropriate external control.

ELIGIBILITY:
Phase 1b Key Inclusion Criteria:

1. Age 21 years or younger at the time of initial ALL diagnosis and age > 1 year at the time of study treatment initiation.
2. Subjects must have a diagnosis of relapsed or refractory ALL with ≥ 5% blasts in the bone marrow (M2 or M3 disease), with or without extramedullary disease.

   -To be eligible, subjects must have had 1 or more prior therapeutic attempts, defined as:
   * Early first relapse (< 36 months from original diagnosis) after achieving a CR (B-ALL) or first relapse any time following the original diagnosis after achieving a CR (T-ALL)
   * First refractory bone marrow relapse occurring any time after original diagnosis after achieving a CR (ie, ≥1 failed attempt to induce a second remission) OR
   * Relapse after achieving a CR following the first or subsequent relapse (i.e., ≥ 2 relapses) OR
   * Failing to achieve a CR from original diagnosis after at least 1 induction attempt
3. Subjects must have fully recovered from the acute toxic effects of all previous chemotherapy, immunotherapy, or radiotherapy treatment before enrollment.
4. Subjects must have a serum creatinine level that is ≤ 1.5 × institutional upper limit of normal (ULN) according to age. If serum creatinine level is > 1.5 × ULN, the subject must have a calculated creatinine clearance or radioisotope glomerular filtration rate (GFR) ≥ 70 mL/min/1.73 m2.
5. Adequate liver function, defined as both of the following:

   * Total bilirubin ≤ 1.5 × institutional ULN except in the presence of Gilbert Syndrome
   * Alanine aminotransferase (ALT) ≤ 5 × institutional ULN
6. Performance status: Karnofsky or Lansky scores ≥ 50 for subjects > 16 years old or ≤ 16 years old, respectively.

Phase 2 Inclusion Criteria:

1. Subject's legally acceptable representative has provided informed consent when the subject is legally too young to provide informed consent and the subject has provided written assent based on local regulations and/or guidelines prior to any study-specific activities/procedures being initiated, except for standard of care local testing as permitted per protocol.
2. Age greater than or equal to 1 month to less than 21 years. Subjects greater than or equal to 18 years must have had their original diagnosis at less than 18 years of age.
3. Subjects must be diagnosed with relapsed or refractory relapsed ALL.
4. Subjects must have a documented first remission, less than 5% blasts in the bone marrow (M1 bone marrow) and no evidence of extramedullary disease.
5. T-cell ALL with bone marrow relapse (defined as greater than or equal to 5% leukemia blasts in bone marrow) or refractory relapse with or without extramedullary disease.

   OR B-cell ALL bone marrow relapse or refractory relapse (defined as greater than or equal to 5% leukemia blasts in bone marrow) after having received a targeted B-cell immune therapy (eg, blinatumomab, inotuzumab or a CAR-T therapy) with or without extramedullary disease..
6. Adequate liver function: bilirubin less than or equal to 1.5 x upper limit of normal (ULN), alanine aminotransferase (ALT) less than or equal to 5 x ULN.
7. Adequate renal function: serum creatinine less than or equal to 1.5 x ULN or glomerular filtration rate (GFR) greater than or equal to 70 mL/min/1.73 m^2; or for children less than 2 years of age, greater than or equal to 50 mL/min/1.73 m^2.
8. Adequate cardiac function: shortening fraction greater than or equal to 30% or ejection fraction greater than or equal to 50%.
9. Karnofsky (subjects greater than or equal to 16 years of age) or Lansky (subjects 12 months to less than 16 years of age) performance status greater than or equal to 50%.
10. Subjects must have fully recovered from the acute toxic effects of all previous chemotherapy, immunotherapy, or radiotherapy treatment before enrollment (for example: recovery from gastrointestinal toxicity may occur more rapidly than less reversible organ toxicities such as sinusoidal obstruction syndrome or non-infectious pneumonitis, for serious prior toxicities recommended discussion with Amgen medical monitor).
11. Life expectancy of greater than 6 weeks per investigator's judgement at time of screening.

Phase 1b Key Exclusion Criteria:

1. Known allergy to any of the drugs used in the study (Subjects who have had a previous allergy to PEG-asparaginase and if able, may receive Erwinia asparaginase at the investigator's discretion)
2. Known allergy to Captisol (a cyclodextrin derivative used to solubilize carfilzomib)
3. Left ventricular fractional shortening < 30%
4. History of ≥ Grade 2 pancreatitis
5. Active graft-versus-host disease requiring systemic treatment
6. Positive culture for or other clinical evidence of infection with bacteria or fungus within 14 days of the initiation of study treatment
7. Down Syndrome
8. Prior therapy restrictions:

   * Subjects must have completed therapy with granulocyte-colony stimulating factor (G-CSF) or other myeloid growth factors at least 7 days before study treatment initiation, or at least 14 days before study treatment initiation, if pegylated myeloid growth factors were administered.
   * Subjects must have completed any type of active immunotherapy (e.g., tumor vaccines) at least 42 days before study treatment initiation.
   * Subjects must have received the last dose of a non-monoclonal antibody biologic agent at least 7 days before study treatment initiation.
   * At least 3 antibody half-lives must have elapsed since the last dose of monoclonal antibody (e.g., 66 days for rituximab and 69 days for epratuzumab) before subjects may initiate study treatment.
   * Subjects must not have received other antineoplastic agents with therapeutic intent, excluding hydroxyurea and antimetabolites administered as part of maintenance chemotherapy, within 7 days prior to study treatment initiation.
9. Hepatitis B infection with positive hepatitis B DNA

Phase 2 Exclusion Criteria:

1. Prior treatment with carfilzomib.
2. Intolerance, hypersensitivity, or inability to receive any of the chemotherapy components of the VXLD regimen. An exception is allowed for allergy to asparaginase products if Erwinia asparaginase is unable to be administered,
3. Autologous HSCT within 6 weeks prior to start of study treatment.
4. Allogeneic HSCT within 3 months prior to start of study treatment.
5. Active GVHD requiring systemic immune suppression.
6. Less than 30 days from discontinuation of immune suppressive therapy administered for the treatment of acute or chronic GVHD.
7. Isolated extramedullary relapse.
8. Positive bacterial or fungal infection within 14 days of enrollment (except for documented line infection, line has been removed, and blood culture after line removal is negative for 5 days prior to first dose of induction therapy). Antibiotics may be administered for prophylaxis as per institutional standards up to and after enrollment.
9. Subjects with less than 3 antibody half-lives since the last dose of monoclonal antibody (eg, 66 days for rituximab, 69 days for epratuzumab, inotuzumab for 36 days), prior to first dose of investigational product must be discussed with the Amgen medical monitor and may be allowed to enroll based on extent of disease or evidence of rapidly rising peripheral or bone marrow blast counts.
10. Cell-based immunotherapy (eg, donor leucocyte infusion, CAR-T cells, tumor vaccines) within 42 days prior to first dose of investigational product. If the Amgen medical monitor agrees, an exception may be granted to the 42-day requirement for subjects with rapidly rising peripheral or bone marrow blast counts.
11. Down's syndrome.
12. Presence of another active cancer.
13. History of grade greater than or equal to 2 pancreatitis within 6 months to screening.
14. Unresolved toxicities from prior anticancer therapy, defined as not having resolved to CTCAE version 4.03 grade 1 or to levels dictated in the eligibility criteria apart from alopecia or toxicities from prior anticancer therapy that are considered irreversible and do not trigger another exclusion criterion (defined as having been present and stable for greater than 4 weeks).
15. Antitumor therapy (chemotherapy, investigational agents, molecular-targeted therapy) within 7 days of day 1 of induction. Exception: hydroxyurea to control peripheral blood leukemic cell counts is allowed until start of investigational product.
16. Active viral infection, including but not limited to cytomegalovirus (CMV), Hepatitis B infection with positive serum hepatitis surface antigen or hepatitis B DNA, HIV, Hepatitis C with detectable hepatitis C RNA. Subjects who have previously received a stem cell transplant must be screened for CMV infection, unless both subject and donor are known to be CMV negative.
17. Currently receiving treatment in another investigational device or product study, or less than 14 days since ending treatment on another investigational device or product study.
18. Uncontrolled arrhythmias or screening ECG with corrected QT interval (QTc) of greater than 470 msec.
19. History or evidence of any other clinically significant disorder, condition or disease (with the exception of those outlined above) that, in the opinion of the investigator or Amgen physician, if consulted, would pose a risk to subject safety or interfere with the study evaluation, procedures or completion.
20. Female subject is pregnant or breastfeeding or planning to become pregnant or breastfeed during treatment and for an additional 6 months after the last dose of any study treatment or for 12 months after last dose of cyclophosphamide if administered during optional consolidation cycle.
21. Female subjects of childbearing potential unwilling to use 1 highly effective method of contraception during treatment and for an additional 6 months after the last dose of any study treatment or for 12 months after last dose of cyclophosphamide if administered during optional consolidation cycle.
22. Female subjects of childbearing potential with a positive pregnancy test assessed at Screening by a serum or urine pregnancy test.
23. Male subjects with a female partner of childbearing potential who are unwilling to practice sexual abstinence (refrain from heterosexual intercourse) or use a condom with spermicide during treatment and for an additional 6 months after the last dose of any study treatment, even if they have undergone a successful vasectomy.
24. Male subjects with a pregnant partner who are unwilling to practice abstinence or use a condom with spermicide during treatment, for duration of pregnancy, and for an additional 6 months after the last dose of any study treatment.
25. Male subjects unwilling to abstain from donating semen or sperm during treatment and for an additional 6 months after the last dose of any study treatment.
26. Known allergy to captisol (a cyclodextrin derivative used to solubilize carfilzomib; for a complete listing of Captisol-enabled drugs, see the Ligand Pharmaceuticals, Inc. website).

Ages: 1 Month to 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 141 (Actual)
Dates: Start 2015-02-16 (Actual); Primary Completion 2024-06-28 (Actual); Study Completion 2024-06-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: MD, Study Director — Amgen
Locations (122):
- United States (22):
  - University of California San Francisco Benioff Childrens Hospital Oakland, Oakland, California
  - Childrens Hospital of Orange County, Orange, California
  - Childrens Hospital Colorado, Aurora, Colorado
  - Childrens Healthcare of Atlanta, Egleston, Atlanta, Georgia
  - Lurie Childrens Hospital of Chicago, Chicago, Illinois
  - The Sidney Kimmel Comprehensive Cancer Center at John Hopkins, Baltimore, Maryland
  - Childrens Hospital and Clinics of Minnesota, Minneapolis, Minnesota
  - Childrens Mercy Hospital, Kansas City, Missouri
  - Rutgers Cancer Institute of New Jersey, New Brunswick, New Jersey
  - Childrens Hospital of New York Presbyterian, New York, New York
  - Levine Childrens Hospital at Carolinas Medical Center d/b/a Atrium Health, Charlotte, North Carolina
  - Cincinnati Childrens Hospital Medical Center, Cincinnati, Ohio
  - The Cleveland Clinic Foundation, Cleveland, Ohio
  - Nationwide Childrens Hospital, Columbus, Ohio
  - Childrens Hospital of Philadelphia, Philadelphia, Pennsylvania
  - Saint Judes Childrens Research Hospital, Memphis, Tennessee
  - Childrens Medical Center, Dallas, Texas
  - Texas Childrens Hospital West Tower, Houston, Texas
  - University of Texas Health Science Center at San Antonio, San Antonio, Texas
  - University of Utah Medical Center Primary Childrens Medical Center, Salt Lake City, Utah
  - West Virginia University Medicine Childrens, Morgantown, West Virginia
  - Medical College of Wisconsin, Milwaukee, Wisconsin
- Argentina (3):
  - Hospital Aleman, Ciudad Autonoma de Buenos Aires, Buenos Aires
  - Hospital Italiano de Buenos Aires, Ciudad Autonoma de Buenos Aires, Buenos Aires
  - Hospital Universitario Austral, Pilar, Buenos Aires
- Australia (5):
  - Sydney Childrens Hospital, Randwick, New South Wales
  - The Childrens Hospital at Westmead, Westmead, New South Wales
  - Queensland Childrens Hospital, South Brisbane, Queensland
  - The Royal Childrens Hospital, Parkville, Victoria
  - Perth Childrens Hospital, Nedlands, Western Australia
- St Anna Kinderspital, Vienna, Austria
- Brazil (11):
  - Hospital São Rafael - IDOR, Salvador, Estado de Bahia
  - Hospital da Crianca de Brasília, Brasília, Federal District
  - Liga Paranaense do Combate ao Cancer - Hospital Erasto Gaertner, Curitba, Paraná
  - Hospital Pequeno Principe, Curitiba, Paraná
  - Instituto de Medicina Integral Professor Fernando Figueira, Recife, Pernambuco
  - Hospital de Clinicas de Porto Alegre, Porto Alegre, Rio Grande do Sul
  - Hospital da Crianca Santo Antonio Irmandade Santa Casa de Misericordia de Porto Alegre, Porto Alegre, Rio Grande do Sul
  - Fundacao Pio 12 Hospital de Amor de Barretos, Barretos, São Paulo
  - Hospital das Clinicas da Faculdade de Medicina de Ribeirao Preto da Universidade de Sao Paulo, Ribeirão Preto, São Paulo
  - Itaci Instituto de Tratamento do Cancer Infantil, São Paulo, São Paulo
  - Beneficencia Portuguesa de Sao Paulo, São Paulo
- University Multiprofile Hospital for Active Treatment Tsaritsa Yoanna-ISUL EAD, Sofia, Bulgaria
- Centre Hospitalier Universitaire Sainte-Justine, Montreal, Quebec, Canada
- Chile (2):
  - Hospital Luis Calvo Mackenna, Santiago
  - Hospital Roberto del Rio, Santiago
- Colombia (2):
  - Sociedad de Oncologia y Hematologia del Cesar, Valledupar, Cesar Department
  - Clinica Imbanaco S.A.S, Cali, Valle del Cauca Department
- Fakultni nemocnice Brno, Brno, Czechia
- University Hospital Rigshospitalet, København Ø, Denmark
- France (6):
  - Centre Hospitalier Universitaire de Bordeaux - Hopital Pellegrin, Bordeaux
  - Centre Hospitalier Regional Universitaire de Lille, Lille
  - Hopital Armand Trousseau, Paris
  - Hopital Robert Debre, Paris
  - Centre Hospitalier Universitaire de Toulouse - Hopital des enfants, Toulouse
  - Centre Hospitalier Universitaire de Nancy - Hopital Enfants de Brabois, Vandœuvre-lès-Nancy
- Greece (5):
  - Agia Sofia Children Hospital, Athens
  - Agia Sofia Children Hospital, Goudi
  - General Children Hospital Panagioti and Aglaias Kyriakou, Goudi
  - General University Hospital of Patras Panagia i Voithia, Pátrai
  - Ippokrateio General Hospital of Thessaloniki, Thessaloniki
- Hong Kong Childrens Hospital, Kowloon Bay, Hong Kong
- Sheba Medical Center, Tel Litwinsky, Israel
- Italy (9):
  - Azienda Ospedaliera Universitaria Consorziale Policlinico di Bari, Bari
  - Azienda Ospedaliera Universitaria Policlinico Vittorio Emanuele Presidio Ospedaliero G Rodolico, Catania
  - IRCCS Istituto Giannina Gaslini, Genova
  - Fondazione IRCCS San Gerardo dei Tintori, Monza (MB)
  - Azienda Ospedaliera di Rilievo Nazionale Santobono Pausilipon, Napoli
  - Azienda Ospedaliera di Padova, Padua
  - Fondazione IRCCS Policlinico San Matteo, Pavia
  - IRCCS Ospedale Pediatrico Bambino Gesu, Roma
  - Azienda Ospedaliera Citta della Salute e della Scienza Torino Ospedale Infantile Regina Margherita, Torino
- Mexico (4):
  - BRCR Global Mexico, Guadalajara, Jalisco
  - BRCR Global Mexico, Mexico City, Mexico City
  - Instituto Nacional de Pediatria, Mexico City, Mexico City
  - BRCR Global Mexico, Puebla City
- Prinses Maxima Centrum voor Kinderoncologie, Utrecht, Netherlands
- Oslo Universitetssykehus Rikshospitalet, Oslo, Norway
- Poland (6):
  - Uniwersytecki Szpital Dzieciecy w Krakowie, Krakow
  - CSK Uniwersytetu Medycznego w Lodzi Uniwersyteckie Centrum Pediatrii im Marii Konopnickiej, Lodz
  - Uniwersytecki szpital dzieciecy, Lublin
  - Uck wum dzieciecy szpital kliniczny im jozefa polikarpa brudzinskiego, Warsaw
  - Uniwersytecki Szpital Kliniczny im Jana Mikulicza-Radeckiego we Wroclawiu, Wroclaw
  - SPSK nr 1 im Prof Stanislawa Szyszko Slaskiego Uniwersytetu Medycznego w Katowicach, Zabrze
- Portugal (3):
  - Centro Hospitalar Universitario de Coimbra, Coimbra
  - Instituto Portugues de Oncologia de Lisboa Francisco Gentil, EPE, Lisbon
  - Instituto Portugues de Oncologia do Porto Francisco Gentil, EPE, Porto
- Romania (3):
  - Institutul Clinic Fundeni, Bucharest
  - Institutul Oncologic Prof Dr Ion Chiricuta Cluj-Napoca, Cluj-Napoca
  - Spitalul Clinic de Urgenta pentru Copii Louis Turcanu Timisoara, Timișoara
- Russia (3):
  - FSBI N N Blokhin Russian Oncology Research Center Ministry of Health of Russian Federation, Moscow
  - FSBI FSCC of pediatric hematology, oncology and immunology n a Dmitry Rogachev, Moscow
  - SBEI of HPE Saint Petersburg State Medical University na academic I P Pavlov of MoH of RF, Saint Petersburg
- King Fahad Medical City, Riyadh, Saudi Arabia
- Singapore (2):
  - National University Hospital, Singapore
  - KK Womens and Childrens Hospital, Singapore
- Chris Hani Baragwanath Hospital, Johannesburg, South Africa
- South Korea (4):
  - Seoul National University Hospital, Seoul
  - Asan Medical Center, Seoul
  - Samsung Medical Center, Seoul
  - Pusan National University Yangsan Hospital, Yangsan-si, Gyeongsangnam-do
- Spain (3):
  - Hospital Sant Joan de Deu, Esplugues de Llobregat, Catalonia
  - Hospital Universitario Infantil Niño Jesus, Madrid
  - Hospital Universitario La Paz, Madrid
- Karolinska Universitetssjukhuset Solna, Solna, Sweden
- Taiwan (3):
  - National Taiwan University Hospital, Taipei
  - Mackay Memorial Hospital Taipei Branch, Taipei
  - Linkou Chang Gung Memorial Hospital, Taoyuan District
- Thailand (4):
  - King Chulalongkorn Memorial Hospital, Bangkok
  - Phramongkutklao Hospital, Bangkok
  - Ramathibodi Hospital, Bangkok
  - Siriraj Hospital, Bangkok
- Turkey (Türkiye) (9):
  - Acibadem Adana Hastanesi, Adana
  - Ankara Universitesi Tip Fakultesi Hastanesi, Ankara
  - Ankara Bilkent Sehir Hastanesi, Ankara
  - Medical Park Antalya Hastanesi, Antalya
  - Bursa Uludag Universitesi Tip Fakultesi, Bursa
  - Medical Park Bahcelievler Hastanesi, Istanbul
  - Medipol Mega Universite Hastanesi, Istanbul
  - Ege Universitesi Tip Fakultesi, Izmir
  - Erciyes Universitesi Tip Fakultesi Mustafa Eraslan ve Fevzi Mercan Cocuk Hastanesi, Kayseri
- The Royal Marsden NHS Foundation Trust, Sutton, United Kingdom

REFERENCES:
- [Derived] Burke MJ, Ziegler DS, Bautista F, Attarbaschi A, Gore L, Locatelli F, M O'Brien M, Pauly M, Kormany WN, Tian S, Morris CL, Baruchel A. Phase 1b study of carfilzomib with induction chemotherapy in pediatric relapsed/refractory acute lymphoblastic leukemia. Pediatr Blood Cancer. 2022 Dec;69(12):e29999. doi: 10.1002/pbc.29999. Epub 2022 Oct 10. PMID 36215217
- See also: AmgenTrials clinical trials website — http://www.amgentrials.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited in Australia, Argentina, Austria, Brazil, Bulgaria, Canada, Chile, Colombia, Czech Republic, Denmark, France, Greece, Hong Kong, Italy, Israel, Mexico, Netherlands, Norway, Poland, Portugal, Romania, Russia, Saudi Arabia, Singapore, South Africa, South Korea, Spain, Sweden, Taiwan, Thailand, Turkey, the UK and the US between February 2015 and June 2024.
Pre-assignment Details: Phase 1b: Participants underwent a 4-week induction and 4-week consolidation cycle, receiving two treatments. Phase 2: After a 7-day screening, participants received VXLD (vincristine, PEG-asparaginase, daunorubicin, dexamethasone) with carfilzomib during a 28-day induction. One B-cell group participant did not receive carfilzomib and was excluded from the primary analysis. Participants were followed for up to 2 years post-treatment.
Groups:
- Phase 1b: Dose Escalation 1 (20 mg/m^2): Participants with relapsed or refractory ALL received carfilzomib 20 mg/m^2 in combination with R3 intravenously (IV) for approximately 9 weeks (1-week lead-in window, 28-day induction cycle, and 28-day optional consolidation cycle).
- Phase 1b: Dose Escalation 1 (20/27 mg/m^2): Participants with relapsed or refractory ALL received carfilzomib 20 mg/m^2 for the first dose, followed by the target 27 mg/m^2 dose in combination with R3 IV for approximately 9 weeks (1-week lead-in window, 28-day induction cycle, and 28-day optional consolidation cycle).
- Phase 1b: Dose Escalation 2 (20/27 mg/m^2): Participants with relapsed or refractory ALL received carfilzomib 20 mg/m^2 for the first dose, followed by the target 27 mg/m^2 dose in combination with VXLD IV for approximately 8 weeks (28-day induction cycle, and 28-day optional consolidation cycle).
- Phase 1b: Dose Escalation 2 (20/36 mg/m^2): Participants with relapsed or refractory ALL received carfilzomib 20 mg/m^2 for the first dose, followed by the target 36 mg/m^2 dose in combination with VXLD IV for approximately 8 weeks (28-day induction cycle, and 28-day optional consolidation cycle).
- Phase 1b: Dose Escalation 2 (20/45 mg/m^2): Participants with relapsed or refractory ALL received carfilzomib 20 mg/m^2 for the first dose, followed by the target 45 mg/m^2 dose in combination VXLD IV for approximately 8 weeks (28-day induction cycle, and 28-day optional consolidation cycle).
- Phase 1b: Dose Escalation 2 (20/56 mg/m^2): Participants with relapsed or refractory ALL received carfilzomib 20 mg/m^2 for the first dose, followed by the target 56 mg/m^2 dose in combination VXLD IV for approximately 8 weeks (28-day induction cycle, and 28-day optional consolidation cycle).
- Phase 2: B-cell (20/56 mg/m^2): Eligible participants with relapsed or refractory ALL (B-cell, after having received a targeted B-cell therapy) were treated with VXLD plus carfilzomib 20/56 mg/m^2 for 1 cycle (induction), followed by assessment of treatment response. Participants who did not show progression during induction underwent a bone marrow and extramedullary disease evaluation after completion of induction therapy. Participants without disease progression after induction could at the investigator's discretion, be treated with 1 28-day consolidation cycle of BFM therapy (cyclophosphamide, cytarabine, 6-mercaptopurine, PEG-asparaginase, vincristine), and IT therapy plus carfilzomib.
- Phase 2: T-cell (20/56 mg/m^2): Eligible participants with relapsed or refractory ALL (T-cell) were treated with VXLD plus carfilzomib 20/56 mg/m^2 for 1 cycle (induction), followed by assessment of treatment response. Participants who did not show progression during induction underwent a bone marrow and extramedullary disease evaluation after completion of induction therapy. Participants without disease progression after induction could at the investigator's discretion, be treated with 1 28-day consolidation cycle of BFM therapy (cyclophosphamide, cytarabine, 6-mercaptopurine, PEG-asparaginase, vincristine), and IT therapy plus carfilzomib.
Period: Overall Study
Arm/Group | Phase 1b: Dose Escalation 1 (20 mg/m^2) | Phase 1b: Dose Escalation 1 (20/27 mg/m^2) | Phase 1b: Dose Escalation 2 (20/27 mg/m^2) | Phase 1b: Dose Escalation 2 (20/36 mg/m^2) | Phase 1b: Dose Escalation 2 (20/45 mg/m^2) | Phase 1b: Dose Escalation 2 (20/56 mg/m^2) | Phase 2: B-cell (20/56 mg/m^2) | Phase 2: T-cell (20/56 mg/m^2)
Started | 5 | 6 | 3 | 7 | 4 | 10 | 62 | 44
Received Carfilzomib During Induction Therapy | 5 | 6 | 3 | 7 | 4 | 10 | 61 | 44
Received Carfilzomib During Consolidation Therapy | 2 | 1 | 1 | 5 | 3 | 3 | 25 | 20
Completed | 5 | 3 | 3 | 7 | 4 | 5 | 19 | 13
Not Completed | 0 | 3 | 0 | 0 | 0 | 5 | 43 | 31
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2
Not completed — Death | 0 | 2 | 0 | 0 | 0 | 3 | 41 | 29
Not completed — Lost to Follow-up | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Not completed — Withdrawal prior to Carfilzomib dosing | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Not completed — Decision by sponsor | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Not completed — Protocol-specified criteria | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Phase 1b: Safety Analysis Set (SAS): All participants who received any amount of the study treatment regimen.
  Phase 2: The baseline population included participants enrolled in 20140106, in the primary analysis set (PAS) who received at least 1 dose of carfilzomib.
Groups:
- Phase 1b: Dose Escalation 1 (20 mg/m^2): Participants with relapsed or refractory ALL received carfilzomib 20 mg/m^2 in combination with R3 IV for approximately 9 weeks (1-week lead-in window, 28-day induction cycle, and 28-day optional consolidation cycle).
- Total: Total of all reporting groups
Arm/Group | Phase 1b: Dose Escalation 1 (20 mg/m^2) | Phase 1b: Dose Escalation 1 (20/27 mg/m^2) | Phase 1b: Dose Escalation 2 (20/27 mg/m^2) | Phase 1b: Dose Escalation 2 (20/36 mg/m^2) | Phase 1b: Dose Escalation 2 (20/45 mg/m^2) | Phase 1b: Dose Escalation 2 (20/56 mg/m^2) | Phase 2: B-cell (20/56 mg/m^2) | Phase 2: T-cell (20/56 mg/m^2) | Total
Number analyzed (Participants) | 5 | 6 | 3 | 7 | 4 | 10 | 61 | 44 | 140
Age, Customized [Count of Participants; unit: Participants]
  < 1 month | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  1 month - <= 17 years | 5 | 6 | 3 | 7 | 3 | 9 | 57 | 41 | 131
  > 17 years | 0 | 0 | 0 | 0 | 1 | 1 | 4 | 3 | 9
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 3 | 0 | 1 | 1 | 3 | 19 | 5 | 35
  Male | 2 | 3 | 3 | 6 | 3 | 7 | 42 | 39 | 105
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 0 | 1 | 2 | 0 | 0 | 28 | 11 | 43
  Not Hispanic or Latino | 4 | 6 | 2 | 5 | 4 | 10 | 33 | 33 | 97
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 2 | 4
  Asian | 0 | 0 | 0 | 0 | 0 | 1 | 9 | 6 | 16
  Black or African American | 0 | 1 | 0 | 0 | 0 | 2 | 2 | 2 | 7
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  White | 5 | 5 | 2 | 7 | 3 | 6 | 38 | 33 | 99
  Other (Indian, Brown, Brazilian indigenous, Hispanic Mestizo, Mestizo breed, Hispanic, and Mixed) | 0 | 0 | 1 | 0 | 1 | 1 | 9 | 1 | 13
  Multiple | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
  Unknown | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Secondary Outcome: Phase 1b: Maximum Concentration (Cmax) of Carfilzomib Alone and in Combination
Description: The PK parameter estimates for carfilzomib were estimated from plasma concentration-time profiles using standard noncompartmental approaches over the complete sampling interval.
Time Frame: Lead-in Cycle Day 1 (7-day cycle) and Induction Cycle Day 8 (28-day cycle): pre-dose, 15 minutes (m) after the start of infusion, immediately (within 2m) before the end of infusion (EOI), EOI, 10m, 30m, 1 hour (h), 2 h, and 4h post-dose
Population: Phase 1b PK Analysis Set: All participants who received the study treatment regimen during the lead-in cycle and induction cycles, and had available data. Phase 1b Dose Escalation 2 arms did not have a 1-week lead-in cycle.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Phase 1b: Dose Escalation 1 (20 mg/m^2) | Phase 1b: Dose Escalation 1 (20/27 mg/m^2) | Phase 1b: Dose Escalation 2 (20/27 mg/m^2) | Phase 1b: Dose Escalation 2 (20/36 mg/m^2) | Phase 1b: Dose Escalation 2 (20/45 mg/m^2) | Phase 1b: Dose Escalation 2 (20/56 mg/m^2)
Number analyzed (Participants) | 5 | 6 | 3 | 6 | 3 | 9
ng/mL
  Dose Escalation 1 - Lead in Cycle Day 1: number analyzed (Participants) | 5 | 6 | 0 | 0 | 0 | 0
  Dose Escalation 1 - Lead in Cycle Day 1 | 927 (259) | 637 (241) |  |  |  |
  Induction cycle Day 8: number analyzed (Participants) | 5 | 4 | 3 | 6 | 3 | 9
  Induction cycle Day 8 | 771 (151) | 792 (580) | 445 (260) | 1070 (359) | 1630 (875) | 11200 (16400)

2. Secondary Outcome: Phase 1b: Area Under the Curve (AUC) From Time 0 to the Last Quantifiable Timepoint (AUClast) of Carfilzomib
Description: as for outcome 1
Time Frame: Lead-in Cycle Day 1 (7-day cycle) and Induction Cycle Day 8 (28-day cycle): pre-dose, 15m after the start of infusion, immediately (within 2m) before the EOI, EOI, 10m, 30m, 1h, 2 h, and 4h post-dose
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: hr*ng/mL
Arm/Group | Phase 1b: Dose Escalation 1 (20 mg/m^2) | Phase 1b: Dose Escalation 1 (20/27 mg/m^2) | Phase 1b: Dose Escalation 2 (20/27 mg/m^2) | Phase 1b: Dose Escalation 2 (20/36 mg/m^2) | Phase 1b: Dose Escalation 2 (20/45 mg/m^2) | Phase 1b: Dose Escalation 2 (20/56 mg/m^2)
Number analyzed (Participants) | 5 | 6 | 3 | 6 | 3 | 9
hr*ng/mL
  Dose Escalation 1 - Lead in Cycle Day 1: number analyzed (Participants) | 5 | 6 | 0 | 0 | 0 | 0
  Dose Escalation 1 - Lead in Cycle Day 1 | 387 (125) | 240 (113) |  |  |  |
  Induction Cycle Day 8: number analyzed (Participants) | 5 | 4 | 3 | 6 | 3 | 9
  Induction Cycle Day 8 | 361 (160) | 374 (273) | 214 (155) | 529 (210) | 829 (479) | 4000 (6370)

3. Secondary Outcome: Phase 1b: AUC From Time 0 to Infinity (AUCinf) of Carfilzomib
Description: as for outcome 1
Time Frame: as for outcome 2
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: hr*ng/ mL
Arm/Group | Phase 1b: Dose Escalation 1 (20 mg/m^2) | Phase 1b: Dose Escalation 1 (20/27 mg/m^2) | Phase 1b: Dose Escalation 2 (20/27 mg/m^2) | Phase 1b: Dose Escalation 2 (20/36 mg/m^2) | Phase 1b: Dose Escalation 2 (20/45 mg/m^2) | Phase 1b: Dose Escalation 2 (20/56 mg/m^2)
Number analyzed (Participants) | 5 | 5 | 1 | 5 | 3 | 5
hr*ng/ mL
  Dose Escalation 1 - Lead in Cycle Day 1: number analyzed (Participants) | 5 | 5 | 0 | 0 | 0 | 0
  Dose Escalation 1 - Lead in Cycle Day 1 | 387 (124) | 268 (101) |  |  |  |
  Induction Cycle Day 8: number analyzed (Participants) | 4 | 4 | 1 | 5 | 3 | 5
  Induction Cycle Day 8 | 368 (184) | 374 (273) | 406 (0.0) | 565 (243) | 848 (510) | 1300 (1440)

4. Secondary Outcome: Phase 1b: Percentage of Participants Who Achieved a Combined CR and CR Without Platelet Recovery (CRp) at the End of Induction Cycle
Description: CR was defined as the attainment of M1 bone marrow status with no evidence of circulating blasts or extramedullary disease and with recovery of peripheral counts (ANC > 750 mcl and platelet count > 75,000 mcl). CRp was defined as the attainment of M1 bone marrow status with no evidence of circulating blasts or extramedullary disease and with recovery of ANCs (ANC > 750 mcl), but with insufficient recovery of platelets (< 75,000 mcl).
Time Frame: Up to approximately Day 29 of Induction Cycle (28-days cycle, assessment on Day 29)
Population: Phase 1b Induction SAS: All participants who received any amount of the study treatment regimen during the induction period and had available data.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Phase 1b: Dose Escalation 1 (20 mg/m^2) | Phase 1b: Dose Escalation 1 (20/27 mg/m^2) | Phase 1b: Dose Escalation 2 (20/27 mg/m^2) | Phase 1b: Dose Escalation 2 (20/36 mg/m^2) | Phase 1b: Dose Escalation 2 (20/45 mg/m^2) | Phase 1b: Dose Escalation 2 (20/56 mg/m^2)
Number analyzed (Participants) | 5 | 5 | 3 | 7 | 4 | 10
Percentage of participants | 40.0 [5.3 to 85.3] | 20.0 [0.5 to 71.6] | 33.3 [0.8 to 90.6] | 28.6 [3.7 to 71.0] | 25.0 [0.6 to 80.6] | 20.0 [2.5 to 55.6]

5. Secondary Outcome: Phase 1b: Percentage of Participants Achieving Minimal Residual Disease (MRD) Status of <10-³ and <10-⁴ Lymphoblasts at the End of Induction Cycle
Description: MRD was defined as the quantification of residual lymphoblast in the blood. Assessed by next generation sequencing (NGS).
Time Frame: Up to approximately Day 29 of Induction Cycle (28-days cycle, assessment on Day29)
Population: as for outcome 4
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Phase 1b: Dose Escalation 1 (20 mg/m^2) | Phase 1b: Dose Escalation 1 (20/27 mg/m^2) | Phase 1b: Dose Escalation 2 (20/27 mg/m^2) | Phase 1b: Dose Escalation 2 (20/36 mg/m^2) | Phase 1b: Dose Escalation 2 (20/45 mg/m^2) | Phase 1b: Dose Escalation 2 (20/56 mg/m^2)
Number analyzed (Participants) | 5 | 5 | 3 | 7 | 4 | 10
Percentage of Participants
  Achieved MRD status < 10^3 lymphoblasts | 0 [NA to NA] — Dispersion was not estimable as 0 participants achieved MRD status | 0 [NA to NA] — Dispersion was not estimable as 0 participants achieved MRD status | 0 [NA to NA] — Dispersion was not estimable as 0 participants achieved MRD status | 14.3 [0.4 to 57.9] | 25.0 [0.6 to 80.6] | 0 [NA to NA] — Dispersion was not estimable as 0 participants achieved MRD status
  Achieved MRD status < 10^4 lymphoblasts | 0 [NA to NA] — Dispersion was not estimable as 0 participants achieved MRD status | 0 [NA to NA] — Dispersion was not estimable as 0 participants achieved MRD status | 0 [NA to NA] — Dispersion was not estimable as 0 participants achieved MRD status | 14.3 [0.4 to 57.9] | 25.0 [0.6 to 80.6] | 0 [NA to NA] — Dispersion was not estimable as 0 participants achieved MRD status

6. Secondary Outcome: Phase 2: Number of Participants Who Experienced TEAEs
Description: An AE is any untoward medical occurrence in a clinical study participant irrespective of a causal relationship with the study treatment. TEAEs are AEs that occurred after the start of study treatment and up to the end of the study or 30 days of the last study treatment, whichever is earlier. Any clinically significant changes in vital signs, electrocardiograms, and clinical laboratory tests that occurred after study treatment administration were recorded as TEAEs. TRAEs were TEAEs considered related to at least one study drug by the investigator, including those with unknown relationship. An SAE was defined as any untoward medical occurrence that resulted in death, was immediately life threatening, required in-patient hospitalization or prolongation of existing hospitalization, resulted in persistent or significant disability/incapacity, a congenital anomaly/birth defect, or another medically important serious event.
Time Frame: From first dose up to 30 days after the last dose of study treatment; maximum duration of treatment was 8 weeks
Population: Phase 2 Safety Analysis Set: All participants enrolled to study 20140106 who received at least 1 dose of carfilzomib.
Measure: Count of Participants; unit: Participants
Arm/Group | Phase 2: B-cell (20/56 mg/m^2) | Phase 2: T-cell (20/56 mg/m^2)
Number analyzed (Participants) | 61 | 44
Participants
  TEAEs | 61 | 44
  SAEs | 44 | 31
  Fatal TEAEs | 15 | 3
  TRAEs | 50 | 39
  Serious TRAEs | 25 | 24
  Fatal TRAEs | 5 | 1

7. Secondary Outcome: Phase 2: Percentage of Participants With CR With Incomplete Hematologic Recovery (CRi) After Induction Therapy or Better Remission Status
Description: CR was defined as: a. Attainment of M1 bone marrow status with no evidence of circulating blasts or extramedullary disease. b. Recovery of peripheral counts: - ANC ≥ 1000/µL - Platelet count ≥ 100 000/µL.
  CRi was defined as:
  1. Attainment of M1 bone marrow status with no evidence of circulating blasts or extramedullary disease
  2. ANC and platelet counts not fulfilling criteria for CR with partial hematologic recovery (CRh), CR without platelet recovery (CRp), or CR.
  CRp was defined as:
  a. Attainment of M1 bone marrow status with no evidence of circulating blasts or extramedullary disease b. Recovery of peripheral counts: i. ANC ≥ 1000/µL ii. Platelet count < 100 000/µL.
  CRh was defined as:
  1. Attainment of M1 bone marrow status with no evidence of circulating blasts or extramedullary disease
  2. Recovery of peripheral counts:
  i. ANC ≥ 500/µL but < 1000/µL ii. Platelet count ≥ 50 000/µL but < 100 000/µL. Data was IPTW adjusted.
Time Frame: Up to Day 50 (28-day cycle of induction therapy + recovery window from Day 29 to Day 45 [up to Day 50 for infants])
Population: Phase 2: Participants enrolled in 20140106, in the PAS, who received at least 1 dose of carfilzomib.
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Phase 2: B-cell (20/56 mg/m^2) | Phase 2: T-cell (20/56 mg/m^2)
Number analyzed (Participants) | 61 | 44
Percentage of Participants | 42.6 [30.2 to 55.0] | 27.3 [14.1 to 40.4]
Statistical Analysis 1: Comparison: Phase 2: B-cell (20/56 mg/m^2) vs Phase 2: T-cell (20/56 mg/m^2); Test type: Other; The objective of this endpoint was to compare the rate of CRi or better status against an external control arm selected from an observational study (Amgen 20180065). The rate of CRi or better status in the external control arm was 26.3% (95% CI: 15.1, 37.5) for B-Cell participants with treatment difference odds ratio of 2.082 (95% CI: 0.968, 4.477). For T-Cell participants the rate of CRi or better status was 18.6% (95% CI: 7.1, 30.0) with treatment difference odds ratio of 1.646 (95% CI: 0.639. 4.245)

8. Secondary Outcome: Phase 2: Event Free Survival (EFS)
Description: EFS was defined as time from initiation of therapy until treatment failure (defined as failure to reach at least a CRi after consolidation or after induction in participants that did not receive consolidation), relapse, or death from any cause. CRi was defined as: a. Attainment of M1 bone marrow status with no evidence of circulating blasts or extramedullary disease b. ANC and platelet counts not fulfilling criteria for CRh, CRp, or CR.
  Data was IPTW adjusted. Medians were estimated using the Kaplan-Meier (KM) method.
Time Frame: Up to approximately 2 years
Population: Phase 2: Participants enrolled in 20140106, in the PAS, who received at least 1 dose of carfilzomib.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Phase 2: B-cell (20/56 mg/m^2) | Phase 2: T-cell (20/56 mg/m^2)
Number analyzed (Participants) | 61 | 44
Months | 1.18 [0.95 to 2.24] | 1.20 [0.95 to 1.48]
Statistical Analysis 1: Comparison: Phase 2: B-cell (20/56 mg/m^2) vs Phase 2: T-cell (20/56 mg/m^2); Test type: Other; The objective of this endpoint was to compare EFS in study 20140106 with EFS in an external control arm selected from an observational study (Amgen 20180065). The median duration in months in the external control arm was 3.62 (95% CI: 1.55, 5.36) for B-cell participants, with a treatment difference hazard ration of 1.435 (95% CI: 0.976, 2.111). For T-Cell participants the median in months was 2.93 (95% CI: 0.95, 5.10) with a treatment difference hazard ratio of 1.404 (95% CI: 0.869, 2.270)

9. Secondary Outcome: Phase 2: Overall Survival (OS)
Description: OS was defined as time from initiation of therapy until death from any cause.
  Data was IPTW adjusted. Medians were estimated using the KM method.
Time Frame: Up to approximately 2 years
Population: Phase 2: Participants enrolled in 20140106, in the PAS, who received at least 1 dose of carfilzomib.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Phase 2: B-cell (20/56 mg/m^2) | Phase 2: T-cell (20/56 mg/m^2)
Number analyzed (Participants) | 61 | 44
Months | 5.23 [2.93 to 9.24] | 4.51 [3.49 to 9.18]
Statistical Analysis 1: Comparison: Phase 2: B-cell (20/56 mg/m^2) vs Phase 2: T-cell (20/56 mg/m^2); Test type: Other; The objective of this endpoint was to compare the OS in study 20140106 with OS in an external control arm selected from an observational study (Amgen 20180065). The median OS in months for the B-Cell participants in the external control arm was 8.59 (95% CI: 5.26, 10.59) with a treatment difference hazard ratio of 1.245 (95% CI: 0.805, 1.927). For the T-Cell participants the median OS in months was 7.04 (95% CI: 7.04, NE) with a treatment difference hazard ratio of 1.040 (95% CI: 0.641, 1.688)

10. Secondary Outcome: Phase 2: Duration of Remission (DOR)
Description: DOR was defined as time from earliest of CR, CRp, CRh, or CRi to relapse or death from any cause. CR was defined as: a. Attainment of M1 bone marrow status with no evidence of circulating blasts or extramedullary disease. b. Recovery of peripheral counts: - ANC ≥ 1000/µL - Platelet count ≥ 100 000/µL. CRi was defined as: a. Attainment of M1 bone marrow status with no evidence of circulating blasts or extramedullary disease b. ANC and platelet counts not fulfilling criteria for CRh, CRp) or CR. CRp was defined as: a. Attainment of M1 bone marrow status with no evidence of circulating blasts or extramedullary disease b. Recovery of peripheral counts: i. ANC ≥ 1000/µL ii. Platelet count < 100 000/µL. CRh was defined as: a. Attainment of M1 bone marrow status with no evidence of circulating blasts or extramedullary disease b. Recovery of peripheral counts: i. ANC ≥ 500/µL but < 1000/µL ii. Platelet count ≥ 50 000/µL but < 100 000/µL.
Time Frame: Up to approximately 2 years
Population: Phase 2: Participants enrolled in 20140106, in the PAS, who received at least 1 dose of carfilzomib. Only participants who achieved CRi or a better remission status were included in the analysis. Data was IPTW adjusted. Medians were estimated using the KM method.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Phase 2: B-cell (20/56 mg/m^2) | Phase 2: T-cell (20/56 mg/m^2)
Number analyzed (Participants) | 26 | 14
Months | 7.55 [3.42 to 22.20] | 9.01 [2.57 to NA] — Upper CI limit not evaluable due to insufficient observations occurring above the median.
Statistical Analysis 1: Comparison: Phase 2: B-cell (20/56 mg/m^2) vs Phase 2: T-cell (20/56 mg/m^2); Test type: Other; The DOR in study 20140106 was estimated relative to the DOR in an external control arm selected from an observational study (Amgen 20180065). The median DOR in months in the external control arm was 8.72 (95% CI: 5.07, 32.24) in B-Cell participants. For T-Cell participants the median DOR in months was 5.82 (95% CI: 1.22, 19.80)

11. Secondary Outcome: Phase 2: Percentage of Participants Achieving MRD Status of <10-³ and <10-⁴ Cells in Participants With CR After Induction Therapy
Description: MRD was defined as the number of leukemia cells that remained in a participant's body after treatment. MRD was measured with next generation sequencing (NGS).
Time Frame: Up to Day 50 (28-day cycle of induction therapy + recovery window from Day 29 to Day 45 [up to Day 50 for infants])
Population: Phase 2 Induction Safety Analysis Set: All participants who started the induction cycle and received at least 1 dose of carfilzomib during the induction period.
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Phase 2: B-cell (20/56 mg/m^2) | Phase 2: T-cell (20/56 mg/m^2)
Number analyzed (Participants) | 61 | 44
Percentage of Participants
  Percentage of Participants Achieving MRD <10-³ Cells | 8.2 [2.7 to 18.1] | 4.5 [0.6 to 15.5]
  Percentage of Participants Achieving MRD <10-⁴ Cells | 3.3 [0.4 to 11.3] | 4.5 [0.6 to 15.5]

12. Secondary Outcome: Phase 2: Percentage of Participants Achieving MRD Status of <10-³ and <10-⁴ Cells in Participants With CRi or Better Status After Induction Therapy
Description: MRD was defined as the number of leukemia cells that remained in a participant's body after treatment. MRD was measured with NGS.
Time Frame: Up to Day 50 (28-day cycle of induction therapy + recovery window from Day 29 to Day 45 [up to Day 50 for infants])
Population: as for outcome 11
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Phase 2: B-cell (20/56 mg/m^2) | Phase 2: T-cell (20/56 mg/m^2)
Number analyzed (Participants) | 61 | 44
Percentage of Participants
  Percentage of Participants Achieving MRD <10-³ Cells | 18.0 [9.4 to 30.0] | 9.1 [2.5 to 21.7]
  Percentage of Participants Achieving MRD <10-⁴ Cells | 9.8 [3.7 to 20.2] | 6.8 [1.4 to 18.7]

13. Secondary Outcome: Phase 2: Percentage of Participants Achieving MRD Status of <10-³ and <10-⁴ Cells in Participants With CRi or Better Status After Consolidation Therapy
Description: as for outcome 12
Time Frame: Up to Day 100 (28-day cycle of induction therapy + recovery window from Day 29 to Day 45 [up to Day 50 for infants] + 28-day cycle of consolidation therapy + + recovery window from Day 29 to Day 45 [up to Day 50 for infants])
Population: Phase 2 Consolidation Safety Analysis Set: All participants who started the consolidation cycle and received at least 1 dose of study treatment during the consolidation period.
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Phase 2: B-cell (20/56 mg/m^2) | Phase 2: T-cell (20/56 mg/m^2)
Number analyzed (Participants) | 25 | 20
Percentage of Participants
  Percentage of Participants Achieving MRD <10-³ Cells | 16.0 [4.5 to 36.1] | 20.0 [5.7 to 43.7]
  Percentage of Participants Achieving MRD <10-⁴ Cells | 16.0 [4.5 to 36.1] | 20.0 [5.7 to 43.7]

14. Secondary Outcome: Phase 2: Percentage of Participants Who Underwent Stem Cell Transplant or Chimeric Antigen Receptor T-cell (CAR-T) Without Intervening Relapse Following Protocol-Specified Therapy
Description: Percentage of participants who successfully underwent stem cell transplant or CAR-T therapy without experiencing a relapse after receiving the protocol-specified treatment.
Time Frame: Up to approximately 2 years
Population: Phase 2: Safety analysis set: All participants who received at least 1 dose of carfilzomib.
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Phase 2: B-cell (20/56 mg/m^2) | Phase 2: T-cell (20/56 mg/m^2)
Number analyzed (Participants) | 61 | 44
Percentage of Participants | 19.7 [10.6 to 31.8] | 27.3 [15.0 to 42.8]

15. Secondary Outcome: Phase 2: Percentage of Participants With CRi or Better Remission Status After Consolidation Therapy
Description: CR was defined as: a. Attainment of M1 bone marrow status with no evidence of circulating blasts or extramedullary disease. b. Recovery of peripheral counts: - ANC ≥ 1000/µL - Platelet count ≥ 100 000/µL.
  CRi was defined as:
  1. Attainment of M1 bone marrow status with no evidence of circulating blasts or extramedullary disease
  2. ANC and platelet counts not fulfilling criteria for CRh, CRp, or CR.
  CRp was defined as:
  a. Attainment of M1 bone marrow status with no evidence of circulating blasts or extramedullary disease b. Recovery of peripheral counts: i. ANC ≥ to 1000/µL ii. Platelet count < 100 000/µL.
  CRh was defined as:
  1. Attainment of M1 bone marrow status with no evidence of circulating blasts or extramedullary disease
  2. Recovery of peripheral counts:
  i. ANC ≥ 500/µL but < 1000/µL ii. Platelet count ≥ 50 000/µL but < 100 000/µL.
  Data was IPTW adjusted.
Time Frame: as for outcome 13
Population: as for outcome 13
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Phase 2: B-cell (20/56 mg/m^2) | Phase 2: T-cell (20/56 mg/m^2)
Number analyzed (Participants) | 25 | 20
Percentage of Participants | 36.0 [18.0 to 57.5] | 50.0 [27.2 to 72.8]

16. Secondary Outcome: Phase 2: AUClast of Carfilzomib
Description: AUClast refers to the total exposure of a drug in the body over time, calculated from the time of administration until the last measurable concentration in the blood.
Time Frame: Day 8 of induction cycle (28-days cycle) and Day 1 of consolidation cycle (28-days cycle)
Population: Phase 2 PK analysis set: All participants who received at least 1 dose of carfilzomib, had 1 PK sample collected and a quantifiable number of observations. Per SAP, analysis was not planned to compare T-cell and B-cell.
Measure: Mean (Standard Deviation); unit: hr*ng/mL
Groups:
- Carfilzomib - Day 8 Induction Cycle: Eligible participants with relapsed or refractory acute lymphoblastic leukemia who had pharmacokinetic (PK) assessments on Day 8 of the induction cycle.
- Carfilzomib - Day 1 Consolidation Cycle: Eligible participants with relapsed or refractory acute lymphoblastic leukemia who had PK assessments on Day 1 of the consolidation cycle.
Arm/Group | Carfilzomib - Day 8 Induction Cycle | Carfilzomib - Day 1 Consolidation Cycle
Number analyzed (Participants) | 83 | 34
hr*ng/mL | 4330 (10300) | 9410 (36200)

17. Secondary Outcome: Phase 2: AUCinf of Carfilzomib
Description: AUCinf represents the total drug exposure over time, extrapolated from the time of administration until the drug is completely eliminated from the body.
Time Frame: Day 8 of induction cycle (28-days cycle) and Day 1 of consolidation cycle (28-days cycle)
Population: as for outcome 16
Measure: Mean (Standard Deviation); unit: hr*ng/mL
Groups:
- Carfilzomib - Day 8 Induction Cycle: Eligible participants with relapsed or refractory acute lymphoblastic leukemia who had PK assessments on Day 8 of the induction cycle.
Arm/Group | Carfilzomib - Day 8 Induction Cycle | Carfilzomib - Day 1 Consolidation Cycle
Number analyzed (Participants) | 46 | 23
hr*ng/mL | 4070 (11000) | 1200 (2480)

18. Secondary Outcome: Phase 2: Cmax of Carfilzomib
Description: Cmax is the maximum concentration of a drug in the bloodstream after administration.
Time Frame: Day 8 of induction cycle (28-days cycle) and Day 1 of consolidation cycle (28-days cycle)
Population: as for outcome 16
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Carfilzomib - Day 8 Induction Cycle | Carfilzomib - Day 1 Consolidation Cycle
Number analyzed (Participants) | 83 | 34
ng/mL | 9590 (27800) | 13800 (44200)

19. Secondary Outcome: Phase 2: Terminal Half-life (t1/2,z) of Carfilzomib
Description: T1/2,z refers to the time required for the plasma concentration of a drug to decrease by half during the final phase of elimination from the body.
Time Frame: Day 8 of induction cycle (28-days cycle) and Day 1 of consolidation cycle (28-days cycle)
Population: as for outcome 16
Measure: Mean (Standard Deviation); unit: hour
Arm/Group | Carfilzomib - Day 8 Induction Cycle | Carfilzomib - Day 1 Consolidation Cycle
Number analyzed (Participants) | 46 | 23
hour | 0.371 (0.162) | 0.332 (0.0894)

20. Primary Outcome: Phase 1b: Number of Participants Who Experienced Treatment-emergent Adverse Events (TEAEs)
Description: An adverse event (AE) is any untoward medical occurrence in a clinical study participant irrespective of a causal relationship with the study treatment. TEAEs are AEs that occurred after the start of study treatment and up to the end of the study or 30 days of the last study treatment, whichever is earlier. Any clinically significant changes in vital signs, electrocardiograms, and clinical laboratory tests that occurred after study treatment administration were recorded as TEAEs. Treatment-related AEs (TRAEs) were TEAEs considered related to at least one study drug by the investigator, including those with unknown relationship. A serious AE (SAE) was defined as any untoward medical occurrence that resulted in death, was immediately life threatening, required in-patient hospitalization or prolongation of existing hospitalization, resulted in persistent or significant disability/incapacity, a congenital anomaly/birth defect, or another medically important serious event.
Time Frame: From first dose up to 30 days after the last dose of study treatment; maximum duration of treatment was 8 weeks
Population: Phase 1b Safety Analysis Set: All participants who received any amount of the study treatment regimen.
Measure: Count of Participants; unit: Participants
Groups:
- Phase 1b: Dose Escalation 2 (20/36 mg/m^2): Participants with relapsed or refractory ALL received carfilzomib 20 mg/m^2 for the first dose, followed by the target 36 mg/m^2 dose in combination VXLD IV for approximately 8 weeks (28-day induction cycle, and 28-day optional consolidation cycle).
- Phase 1b: Dose Escalation 2 (20/45 mg/m^2: Participants with relapsed or refractory ALL received carfilzomib 20 mg/m^2 for the first dose, followed by the target 45 mg/m^2 dose in combination VXLD IV for approximately 8 weeks (28-day induction cycle, and 28-day optional consolidation cycle).
Arm/Group | Phase 1b: Dose Escalation 1 (20 mg/m^2) | Phase 1b: Dose Escalation 1 (20/27 mg/m^2) | Phase 1b: Dose Escalation 2 (20/27 mg/m^2) | Phase 1b: Dose Escalation 2 (20/36 mg/m^2) | Phase 1b: Dose Escalation 2 (20/45 mg/m^2 | Phase 1b: Dose Escalation 2 (20/56 mg/m^2)
Number analyzed (Participants) | 5 | 6 | 3 | 7 | 4 | 10
Participants
  All TEAEs | 5 | 6 | 3 | 7 | 4 | 9
  All fatal TEAEs | 0 | 2 | 0 | 0 | 0 | 3
  All TRAEs | 5 | 4 | 3 | 7 | 4 | 8
  All fatal TRAEs | 0 | 0 | 0 | 0 | 0 | 1
  All SAEs | 4 | 4 | 3 | 6 | 4 | 7

21. Primary Outcome: Phase 1b: Number of Participants Who Experienced Dose Limiting Toxicities (DLTs)
Description: A DLT was defined as any of the following toxicities assessed by the investigator as possibly, probably, or definitely attributable to carfilzomib, with protocol defined exclusions: Any Grade 4 nonhematologic toxicity, ≥ Grade 4 neutropenia or ≥ Grade 3 thrombocytopenia.
Time Frame: Up to approximately 35 days
Population: Phase 1b DLT Evaluable Analysis Set: All participants who received all planned dose of carfilzomib and the chemotherapy backbone per protocol during the lead-in window and induction cycle, or received at least one dose of carfilzomib and the chemotherapy backbone per protocol and experienced a DLT prior to completion of the lead-in window or induction cycle, or as clinically indicated.
Measure: Count of Participants; unit: Participants
Arm/Group | Phase 1b: Dose Escalation 1 (20 mg/m^2) | Phase 1b: Dose Escalation 1 (20/27 mg/m^2) | Phase 1b: Dose Escalation 2 (20/27 mg/m^2) | Phase 1b: Dose Escalation 2 (20/36 mg/m^2) | Phase 1b: Dose Escalation 2 (20/45 mg/m^2) | Phase 1b: Dose Escalation 2 (20/56 mg/m^2)
Number analyzed (Participants) | 4 | 4 | 2 | 4 | 3 | 8
Participants
  Haemolytic uraemic syndrome | 0 | 1 | 0 | 0 | 0 | 0
  Platelet count decreased | 0 | 0 | 0 | 0 | 0 | 1
  Pulmonary haemorrhage | 0 | 0 | 0 | 0 | 0 | 1

22. Primary Outcome: Phase 2: Percentage of Participants With Complete Remission (CR) After Induction Therapy
Description: CR was defined as:
  1. Attainment of M1 bone marrow status (less than 5% blasts in a bone marrow aspirate and at least 200 cells counted) with no evidence of circulating blasts or extramedullary disease.
  2. Recovery of peripheral counts:
     * Absolute neutrophil count (ANC) greater than or equal to 1000/µL
     * Platelet count greater than or equal to 100000/µL.
     * Assessed between days 29 and 45
  Data was adjusted as inverse probability of treatment weight (IPTW) for the average treatment effect of the treated (IPTW-ATTW).
Time Frame: Up to Day 50 (28-day cycle of induction therapy + recovery window from Day 29 to Day 45 [Day 36 to Day 50 for infants])
Population: Phase 2: Participants enrolled in 20140106, in the PAS, who received at least 1 dose of carfilzomib.
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Phase 2: B-cell (20/56 mg/m^2) | Phase 2: T-cell (20/56 mg/m^2)
Number analyzed (Participants) | 61 | 44
Percentage of Participants | 14.8 [5.9 to 23.7] | 13.6 [3.5 to 23.8]
Statistical Analysis 1: Comparison: Phase 2: B-cell (20/56 mg/m^2) vs Phase 2: T-cell (20/56 mg/m^2); Test type: Other; The primary objective of this endpoint was to compare the percentage of participants achieving CR after the end of induction therapy in study 20140106 with the percentage of participants achieving CR in an external control arm selected from an observational study (Amgen 20180065). In the external control arm, 7.8% of B-Cell participants (95% confidence interval [CI]: 1.0%, 14.7%) achieved CR, with a treatment difference odds ratio of 2.04 (95% CI: 0.54, 7.66). For T-Cell participants, 9.1% (95% CI: 0.7%, 17.5%) achieved CR, with an odds ratio of 1.58 (95% CI: 0.47, 5.31)

ADVERSE EVENTS:
Time Frame: Phase 1b/2: For deaths, up to approximately 2 years. For TEAEs, from first dose up to 30 days after the last dose of study treatment; maximum duration of treatment was 8 weeks
Description: Serious adverse events and other adverse events are reported for all participants who received at least one dose of study drug. All-cause mortality is reported for all participants enrolled in the study. The MedDRA version is 23.1 for Phase 1b, and 27.0 for Phase 2.
Arm/Group | Phase 1b: Dose Escalation 1 (20 mg/m^2) | Phase 1b: Dose Escalation 1 (20/27 mg/m^2) | Phase 1b: Dose Escalation 2 (20/27 mg/m^2) | Phase 1b: Dose Escalation 2 (20/36 mg/m^2) | Phase 1b: Dose Escalation 2 (20/45 mg/m^2 | Phase 1b: Dose Escalation 2 (20/56 mg/m^2) | Phase 2: B-cell (20/56 mg/m^2) | Phase 2: T-cell (20/56 mg/m^2)
All-Cause Mortality (participants affected / at risk) | 0/5 | 2/6 | 0/3 | 0/7 | 0/4 | 3/10 | 41/62 | 29/44
Serious Adverse Events (participants affected / at risk) | 4/5 | 4/6 | 3/3 | 6/7 | 4/4 | 7/10 | 44/61 | 31/44
Other Adverse Events (participants affected / at risk) | 5/5 | 6/6 | 3/3 | 7/7 | 4/4 | 9/10 | 61/61 | 43/44
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Phase 1b: Dose Escalation 1 (20 mg/m^2) (N=5) | Phase 1b: Dose Escalation 1 (20/27 mg/m^2) (N=6) | Phase 1b: Dose Escalation 2 (20/27 mg/m^2) (N=3) | Phase 1b: Dose Escalation 2 (20/36 mg/m^2) (N=7) | Phase 1b: Dose Escalation 2 (20/45 mg/m^2 (N=4) | Phase 1b: Dose Escalation 2 (20/56 mg/m^2) (N=10) | Phase 2: B-cell (20/56 mg/m^2) (N=61) | Phase 2: T-cell (20/56 mg/m^2) (N=44)
Anaemia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1
Febrile neutropenia (Blood and lymphatic system disorders) | 3 | 2 | 1 | 3 | 1 | 1 | 8 | 3
Hyperleukocytosis (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Leukopenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3
Neutropenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Pancytopenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 4
Angina pectoris (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Cardiac dysfunction (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Tachycardia (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0
Toxic cardiomyopathy (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0
Colitis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Neutropenic colitis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 0
Pancreatitis (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 1
Pancreatitis acute (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 1 | 0 | 1 | 1
Stomatitis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Malaise (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Multiple organ dysfunction syndrome (General disorders) | 0 | 1 | 0 | 0 | 0 | 1 | 1 | 0
Pyrexia (General disorders) | 0 | 0 | 1 | 1 | 0 | 0 | 1 | 3
Cholecystitis acute (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Hepatitis acute (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Hepatobiliary disease (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Alpha haemolytic streptococcal infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Appendicitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Bacteraemia (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Bacterial infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2
Bacterial sepsis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Bronchopulmonary aspergillosis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 1
COVID-19 (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
COVID-19 pneumonia (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Clostridium difficile infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Device related infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Encephalitis (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Escherichia sepsis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 3
Fungaemia (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Fungal infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 2 | 0
Gastroenteritis rotavirus (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Herpes simplex reactivation (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Lower respiratory tract infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Meningitis bacterial (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Necrotising fasciitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Neutropenic sepsis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Pneumonia (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 1 | 4 | 2
Pneumonia fungal (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 1
Pneumonia klebsiella (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Pseudomonal sepsis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Sepsis (Infections and infestations) | 1 | 2 | 0 | 0 | 1 | 0 | 4 | 0
Sepsis syndrome (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Septic shock (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 9 | 2
Severe acute respiratory syndrome (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Soft tissue infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Vascular device infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Viral infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Procedural nausea (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Transfusion reaction (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Aspartate aminotransferase increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Blood creatinine increased (Investigations) | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Body temperature increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
N-terminal prohormone brain natriuretic peptide increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Neutrophil count decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Oxygen saturation decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Dehydration (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Hypoalbuminaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Hypocalcaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 2
Hypomagnesaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Hypophosphataemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Tumour lysis syndrome (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 2 | 2
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2
Cerebral haemorrhage (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Cerebral small vessel ischaemic disease (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Cerebrovascular accident (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Cerebrovascular disorder (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Cognitive disorder (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Consciousness fluctuating (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Encephalopathy (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0
Nervous system disorder (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Peripheral motor neuropathy (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Peripheral sensorimotor neuropathy (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Petit mal epilepsy (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Posterior reversible encephalopathy syndrome (Nervous system disorders) | 0 | 0 | 0 | 3 | 0 | 0 | 1 | 4
Seizure (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Toxic encephalopathy (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Acute kidney injury (Renal and urinary disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Haematuria (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Mediastinal disorder (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Pulmonary alveolar haemorrhage (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Pulmonary haemorrhage (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Pulmonary veno-occlusive disease (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Respiratory disorder (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0
Tachypnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Hypotension (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Hypovolaemic shock (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Jugular vein thrombosis (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Haemolytic uraemic syndrome (Blood and lymphatic system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Enterocolitis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Mucosal inflammation (General disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Hepatic failure (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Drug hypersensitivity (Immune system disorders) | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0
Bacillus bacteraemia (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0
Fusobacterium infection (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Infection in an immunocompromised host (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Pneumonia viral (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Staphylococcal bacteraemia (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Stomatococcal infection (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Systemic candida (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Catheter culture positive (Investigations) | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0
Platelet count decreased (Investigations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Acute lymphocytic leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Brain oedema (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Clonic convulsion (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Dysarthria (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Hydrocephalus (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Neuralgia (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Somnolence (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Confusional state (Psychiatric disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Dyspnoea at rest (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Phase 1b: Dose Escalation 1 (20 mg/m^2) (N=5) | Phase 1b: Dose Escalation 1 (20/27 mg/m^2) (N=6) | Phase 1b: Dose Escalation 2 (20/27 mg/m^2) (N=3) | Phase 1b: Dose Escalation 2 (20/36 mg/m^2) (N=7) | Phase 1b: Dose Escalation 2 (20/45 mg/m^2 (N=4) | Phase 1b: Dose Escalation 2 (20/56 mg/m^2) (N=10) | Phase 2: B-cell (20/56 mg/m^2) (N=61) | Phase 2: T-cell (20/56 mg/m^2) (N=44)
Anaemia (Blood and lymphatic system disorders) | 4 | 5 | 2 | 4 | 3 | 3 | 37 | 23
Febrile neutropenia (Blood and lymphatic system disorders) | 1 | 1 | 1 | 0 | 1 | 3 | 17 | 11
Leukopenia (Blood and lymphatic system disorders) | 0 | 1 | 0 | 0 | 1 | 0 | 12 | 10
Lymphopenia (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 6 | 4
Neutropenia (Blood and lymphatic system disorders) | 2 | 3 | 0 | 1 | 1 | 0 | 24 | 17
Thrombocytopenia (Blood and lymphatic system disorders) | 2 | 1 | 1 | 1 | 0 | 0 | 23 | 20
Tachycardia (Cardiac disorders) | 0 | 2 | 0 | 1 | 3 | 0 | 4 | 0
Abdominal pain (Gastrointestinal disorders) | 1 | 2 | 1 | 2 | 1 | 1 | 9 | 7
Abdominal pain upper (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 3 | 4
Constipation (Gastrointestinal disorders) | 0 | 1 | 1 | 2 | 2 | 1 | 7 | 9
Diarrhoea (Gastrointestinal disorders) | 3 | 2 | 1 | 4 | 0 | 3 | 13 | 9
Nausea (Gastrointestinal disorders) | 4 | 0 | 2 | 5 | 2 | 0 | 8 | 11
Oral pain (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 3
Stomatitis (Gastrointestinal disorders) | 0 | 1 | 0 | 3 | 0 | 0 | 4 | 7
Vomiting (Gastrointestinal disorders) | 4 | 2 | 1 | 2 | 3 | 2 | 7 | 7
Face oedema (General disorders) | 1 | 0 | 0 | 0 | 1 | 0 | 1 | 4
Mucosal inflammation (General disorders) | 0 | 2 | 1 | 0 | 1 | 1 | 5 | 0
Pain (General disorders) | 0 | 0 | 0 | 1 | 0 | 1 | 3 | 7
Pyrexia (General disorders) | 2 | 4 | 2 | 3 | 2 | 3 | 27 | 23
Hyperbilirubinaemia (Hepatobiliary disorders) | 0 | 1 | 0 | 0 | 0 | 1 | 2 | 4
Hypogammaglobulinaemia (Immune system disorders) | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 3
Bacteraemia (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 4 | 0
COVID-19 (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 4 | 3
Pneumonia (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 4 | 3
Rhinovirus infection (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 1 | 4 | 0
Sepsis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 2 | 3
Alanine aminotransferase increased (Investigations) | 3 | 3 | 1 | 3 | 1 | 2 | 21 | 14
Antithrombin III decreased (Investigations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 5
Aspartate aminotransferase increased (Investigations) | 2 | 2 | 0 | 3 | 1 | 0 | 18 | 10
Blood bilirubin increased (Investigations) | 2 | 1 | 1 | 1 | 1 | 0 | 6 | 4
Gamma-glutamyltransferase increased (Investigations) | 1 | 1 | 0 | 1 | 1 | 0 | 7 | 5
International normalised ratio increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 3
Lymphocyte count decreased (Investigations) | 2 | 1 | 0 | 1 | 0 | 1 | 4 | 0
Neutrophil count decreased (Investigations) | 2 | 1 | 1 | 2 | 1 | 1 | 6 | 4
Platelet count decreased (Investigations) | 2 | 2 | 1 | 3 | 2 | 4 | 11 | 4
White blood cell count decreased (Investigations) | 2 | 1 | 1 | 2 | 1 | 0 | 11 | 5
Hyperglycaemia (Metabolism and nutrition disorders) | 3 | 3 | 1 | 0 | 0 | 1 | 3 | 6
Hyperkalaemia (Metabolism and nutrition disorders) | 2 | 2 | 0 | 1 | 0 | 0 | 5 | 1
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 4
Hyperuricaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 8 | 1
Hypoalbuminaemia (Metabolism and nutrition disorders) | 3 | 3 | 1 | 2 | 1 | 1 | 18 | 8
Hypocalcaemia (Metabolism and nutrition disorders) | 2 | 3 | 1 | 1 | 0 | 0 | 11 | 5
Hypoglycaemia (Metabolism and nutrition disorders) | 1 | 3 | 0 | 2 | 0 | 2 | 3 | 3
Hypokalaemia (Metabolism and nutrition disorders) | 3 | 3 | 1 | 3 | 2 | 3 | 15 | 17
Hypomagnesaemia (Metabolism and nutrition disorders) | 2 | 3 | 0 | 0 | 2 | 1 | 5 | 5
Hyponatraemia (Metabolism and nutrition disorders) | 2 | 3 | 1 | 1 | 0 | 2 | 6 | 4
Hypophosphataemia (Metabolism and nutrition disorders) | 3 | 2 | 0 | 1 | 1 | 3 | 5 | 5
Tumour lysis syndrome (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 5 | 2
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 | 0 | 0 | 0 | 0 | 1 | 2 | 3
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 2 | 2 | 0 | 0 | 1 | 4
Pain in extremity (Musculoskeletal and connective tissue disorders) | 2 | 2 | 0 | 4 | 2 | 1 | 4 | 3
Headache (Nervous system disorders) | 2 | 0 | 1 | 3 | 2 | 2 | 8 | 10
Neuropathy peripheral (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 4 | 3
Acute kidney injury (Renal and urinary disorders) | 2 | 0 | 0 | 0 | 0 | 1 | 5 | 2
Haematuria (Renal and urinary disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 3
Cough (Respiratory, thoracic and mediastinal disorders) | 2 | 2 | 1 | 2 | 0 | 0 | 3 | 4
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 2 | 0 | 0 | 2 | 4
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1 | 0 | 0 | 1 | 1 | 4
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 5 | 3
Rash (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 1 | 0 | 4 | 0
Hypertension (Vascular disorders) | 2 | 3 | 1 | 6 | 2 | 7 | 25 | 13
Hypotension (Vascular disorders) | 1 | 0 | 0 | 0 | 3 | 2 | 3 | 4
Bone marrow failure (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1
Coagulopathy (Blood and lymphatic system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 2 | 0
Myelosuppression (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Atrioventricular block (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Bradycardia (Cardiac disorders) | 2 | 0 | 0 | 0 | 1 | 1 | 1 | 2
Cardiac failure (Cardiac disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0
Sinus bradycardia (Cardiac disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 2 | 2
Sinus tachycardia (Cardiac disorders) | 1 | 0 | 0 | 2 | 2 | 1 | 2 | 0
Adrenal insufficiency (Endocrine disorders) | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 1
Cushingoid (Endocrine disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Inappropriate antidiuretic hormone secretion (Endocrine disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1
Diplopia (Eye disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Dry eye (Eye disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Eye irritation (Eye disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Eye pain (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Periorbital oedema (Eye disorders) | 1 | 0 | 0 | 0 | 0 | 1 | 1 | 0
Periorbital swelling (Eye disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Photophobia (Eye disorders) | 1 | 0 | 2 | 0 | 0 | 0 | 0 | 1
Vision blurred (Eye disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0
Abdominal distension (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 3 | 0
Anal fissure (Gastrointestinal disorders) | 0 | 0 | 1 | 1 | 0 | 1 | 3 | 1
Colitis (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 2 | 1
Dental caries (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Dry mouth (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Dyspepsia (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 2 | 0 | 0 | 0
Haematochezia (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 1
Impaired gastric emptying (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Lip dry (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0
Oral mucosal erythema (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Pancreatitis (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 2
Toothache (Gastrointestinal disorders) | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 2 | 0
Catheter site erythema (General disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Catheter site pain (General disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Chills (General disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Fatigue (General disorders) | 2 | 1 | 1 | 1 | 2 | 3 | 1 | 0
Influenza like illness (General disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Multiple organ dysfunction syndrome (General disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Oedema (General disorders) | 1 | 0 | 0 | 2 | 0 | 1 | 1 | 1
Oedema peripheral (General disorders) | 1 | 0 | 0 | 1 | 1 | 0 | 2 | 1
Peripheral swelling (General disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Cholangitis (Hepatobiliary disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Cholecystitis (Hepatobiliary disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Hepatic lesion (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Drug hypersensitivity (Immune system disorders) | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 1
Hypersensitivity (Immune system disorders) | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 1
Immunodeficiency common variable (Immune system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Appendicitis perforated (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Aspergillus infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
Bacterial infection (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Cytomegalovirus infection (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0
Device related bacteraemia (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Device related infection (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 2 | 0
Enterocolitis infectious (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Fungal sepsis (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1
Infection (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Infection in an immunocompromised host (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Oral candidiasis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 2
Oral herpes (Infections and infestations) | 0 | 0 | 1 | 1 | 0 | 0 | 3 | 1
Paronychia (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Pseudomembranous colitis (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0
Septic shock (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Sinusitis (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 3 | 0
Staphylococcal bacteraemia (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1
Stomatococcal infection (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Upper respiratory tract infection (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 1
Varicella zoster virus infection (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Viral upper respiratory tract infection (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Contusion (Injury, poisoning and procedural complications) | 1 | 1 | 0 | 1 | 1 | 0 | 1 | 1
Foreign body ingestion (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Infusion related reaction (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 1
Procedural nausea (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Scratch (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Activated partial thromboplastin time prolonged (Investigations) | 1 | 0 | 0 | 2 | 0 | 0 | 0 | 0
Ammonia (Investigations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Amylase increased (Investigations) | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 1
Aspartate aminotransferase decreased (Investigations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Bacterial test positive (Investigations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Bilirubin conjugated increased (Investigations) | 0 | 0 | 1 | 0 | 1 | 0 | 1 | 1
Blood creatine increased (Investigations) | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 1
Blood creatinine increased (Investigations) | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 2
Blood fibrinogen decreased (Investigations) | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 2
Blood urea increased (Investigations) | 1 | 1 | 0 | 0 | 0 | 0 | 2 | 1
Breath sounds abnormal (Investigations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
C-reactive protein increased (Investigations) | 0 | 0 | 0 | 1 | 0 | 0 | 2 | 2
Candida test positive (Investigations) | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0
Electrocardiogram QT prolonged (Investigations) | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0
Immunoglobulins decreased (Investigations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1
Lipase increased (Investigations) | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 2
Lymphocyte count (Investigations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Protein total abnormal (Investigations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Staphylococcus test positive (Investigations) | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0
Urine protein/creatinine ratio increased (Investigations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Weight decreased (Investigations) | 2 | 2 | 0 | 1 | 1 | 1 | 0 | 1
Weight increased (Investigations) | 2 | 0 | 1 | 0 | 1 | 1 | 1 | 2
Acidosis (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Decreased appetite (Metabolism and nutrition disorders) | 4 | 0 | 1 | 1 | 1 | 0 | 3 | 0
Diabetes mellitus (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Fluid overload (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Hypercalcaemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hypermagnesaemia (Metabolism and nutrition disorders) | 1 | 1 | 0 | 1 | 0 | 0 | 0 | 0
Hypernatraemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 1 | 0 | 1 | 0
Hyperphosphataemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 3 | 2
Vitamin D deficiency (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Bone pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 1
Joint range of motion decreased (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Joint swelling (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Limb discomfort (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0 | 1 | 2 | 1
Neck pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0
Osteonecrosis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Pain in jaw (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 2 | 1
Chloroma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Dizziness (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Epilepsy (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0
Lethargy (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Loss of consciousness (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Neuralgia (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 2
Paraesthesia (Nervous system disorders) | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0
Peripheral motor neuropathy (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Peripheral sensory neuropathy (Nervous system disorders) | 0 | 0 | 0 | 1 | 1 | 1 | 0 | 0
Seizure (Nervous system disorders) | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0
Somnolence (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Syncope (Nervous system disorders) | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0
Abnormal behaviour (Psychiatric disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Affective disorder (Psychiatric disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Agitation (Psychiatric disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0
Anxiety (Psychiatric disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 1
Depression (Psychiatric disorders) | 1 | 0 | 1 | 0 | 0 | 0 | 2 | 1
Insomnia (Psychiatric disorders) | 0 | 1 | 0 | 1 | 2 | 0 | 1 | 2
Irritability (Psychiatric disorders) | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0
Suicidal ideation (Psychiatric disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Chromaturia (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Proteinuria (Renal and urinary disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Renal failure (Renal and urinary disorders) | 0 | 1 | 0 | 0 | 0 | 1 | 1 | 0
Urinary incontinence (Renal and urinary disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Breast pain (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Aspiration (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Dry throat (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Dyspnoea at rest (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 1 | 1 | 0
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 1 | 0 | 0 | 1 | 2
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 2
Pulmonary haemorrhage (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 2 | 1 | 2
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Tachypnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Alopecia (Skin and subcutaneous tissue disorders) | 2 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Dermatitis acneiform (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Dermatitis bullous (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Dermatitis diaper (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Erythema (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 1 | 0 | 1 | 2
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Palmar-plantar erythrodysaesthesia syndrome (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Papule (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Petechiae (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 1 | 3 | 1 | 1
Pruritus (Skin and subcutaneous tissue disorders) | 1 | 0 | 1 | 1 | 1 | 1 | 0 | 0
Purpura (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 2 | 0 | 0 | 0 | 0
Skin lesion (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0
Urticaria (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 1
Flushing (Vascular disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Haematoma (Vascular disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1
Thrombophlebitis (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Clinical Trial Agreement generally does not restrict an investigator's discussion of trial results after completion. The Agreement permits Amgen a limited period of time to review material discussing trial results (typically up to 45 days and possible extension). Amgen may remove confidential information, but authors have final control and approval of publication content. For multicenter studies, the investigator agrees not to publish any results before the first multi-center publication.

DOCUMENTS (2):
  • Study Protocol (2023-08-28): https://cdn.clinicaltrials.gov/large-docs/21/NCT02303821/Prot_000.pdf
  • Statistical Analysis Plan (2023-08-29): https://cdn.clinicaltrials.gov/large-docs/21/NCT02303821/SAP_001.pdf